CLINICAL TRIAL: NCT06489119
Title: Single-cell Multi-omics Analyses of OCT-diagnosed Plaque Subtypes in Coronary Artery Disease - a Prospective, Observational Study
Brief Title: Single-cell Multi-omics Analyses of OCT-diagnosed Plaque Subtypes in Coronary Artery Disease (MOOP-CAD)
Acronym: MOOP-CAD
Status: Recruiting | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director of Department of Cardiology, Harbin Medical University
Other Study IDs: KY2024-084
Record Dates: First submitted 2024-06-17; First posted 2024-07-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary atherosclerosis; Optical coherence tomography; Multi-omics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control group: Patients with angiographic diameter stenosis <20%
- Stable plaque group: Angiographic diameter stenosis >50% with no TCFA lesions in the most severely narrowed native coronary artery (target vessel).
- Vulnerable plaque group: Angiographic diameter stenosis >50% with TCFA lesions in the most severely narrowed native coronary artery (target vessel).
- Plaque rupture group: Patient diagnosed as AMI with plaque rupture detected by OCT.
- Plaque erosion group: Patient diagnosed as AMI with plaque erosion detected by OCT.

SUMMARY:
The MOOP-CAD study program characterizes, for the first time, the pathophysiological processes and molecular mechanisms of coronary atherosclerotic plaque progression by combining in vivo intravascular imaging techniques with circulating immune single-cell multi-omics analysis. In this study, the investigators evaluate the imaging characteristics of coronary plaques by optical coherence tomography (OCT) and invasive angiography, and study the correlation between plaque characteristics and the multi-omics immune characteristic profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age ≥ 18 years and ≤ 85 years.
2. Ability to understand the requirements of the study and to provide informed consent.

Control group:

Patients with coronary angiographic diameter stenosis <20%.

Stable plaque group:

1. Have been clinically stable for at least 6 months.
2. Presence of ≥1 lesion with angiographic diameter stenosis >50% with no TCFA lesions in the most severely narrowed native coronary artery (target vessel). TCFA was defined as a lipidic plaque with the thinnest FCT <75 mm and maximum lipid arc >180°.
3. Rule out elevation of troponin or myocardial enzymology.

Vulnerable plaque group:

1. Have been clinically stable for at least 6 months.
2. Presence of ≥1 lesion with angiographic diameter stenosis >50% with TCFA lesions in the most severely narrowed native coronary artery (target vessel).
3. Rule out elevation of troponin or myocardial enzymology.

Plaque rupture group:

1. Persistent chest pain for 30 minutes, arrival at the hospital within 24 hours from symptom onset. ST-segment elevation of >0.1 mV in ≥2 contiguous leads or new-onset left bundle branch block, and high sensitive Troponin T or I or CK/CK-MB above upper reference value.
2. Exist clearly identified culprit lesion.
3. Plaque rupture was defined by the presence of a discontinuity of the fibrous cap with a cavity formed inside the plaque.

Plaque erosion group:

1. Persistent chest pain for 30 minutes, arrival at the hospital within 24 hours from symptom onset. ST-segment elevation of >0.1 mV in ≥2 contiguous leads or new-onset left bundle branch block, and high sensitive Troponin T or I or CK/CK-MB above upper reference value.
2. Exist clearly identified culprit lesion.
3. Plaque erosion was defined by the presence of the attached thrombus overlying the intact fibrous cap of the atherosclerotic plaque, luminal surface irregularity at the culprit lesion in the absence of thrombus, or attenuation of the underlying plaque by thrombus without superficial lipid or calcium at the site of the thrombus.

Exclusion Criteria:

1. Cardiogenic shock or circulatory depression，life-threatening arrhythmia.
2. Known systolic heart failure with LVEF ≤30%.
3. Severe systemic diseases (end-stage renal disease, serious liver dysfunction, chronic active inflammatory diseases, active oncologic diseases, autoimmune diseases).
4. Septicemia, acute inflammatory event with fever.
5. Patients with organ transplants or patients on the waiting list for an organ transplant.
6. Previous CABG treatment, PCI treatment of the target vessel, and PCI treatment of non-target vessels within 1 year.
7. Thrombolysis before PCI.
8. Stenosis of the left main artery ≥50%.
9. Characteristics rendering high-quality OCT imaging unlikely such as chronic total occlusion, pronounced tortuosity, heavily calcified vessels.
10. Infarcted vessel with a diameter >4mm or <2.5mm.
11. "No-reflow" (TIMI 0-1) after thrombus aspiration or predilatation.
12. Other subjects deemed unsuitable for study by investigators.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who meet the preset inclusion criteria for each group of people, understand the research requirements and treatment procedures, and sign the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE | 1 year following hospital discharge
  The incidence of major adverse cardiovascular events in patients (Major adverse cardiovascular events is defined as the composite of all-cause death, recurrent myocardial infarction, revascularization, unplanned readmission for angina exacerbation or unstable angina)

SECONDARY OUTCOMES:
Incidence of SCD | 1 year following hospital discharge
  The incidence of sudden cardiac death in patients
Incidence of nonfatal myocardial infarction | 1 year following hospital discharge
  The incidence of nonfatal myocardial infarction in patients
Incidence of target vessel revascularization | 1 year following hospital discharge
  The incidence of target vessel revascularization in patients

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - China-Japan Union Hospital of Jilin, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No